CLINICAL TRIAL: NCT03417206
Title: Comparative Study of Influence of Total Intravenous Anaesthesia (TIVA) and Volatile Anaesthesia Using Sevoflurane or Desflurane on the Intraoperative Blood Loss During Functional Endoscopic Sinus Surgery
Brief Title: PRD-guided Analgesia During FESS for Intraoperative Blood Loss
Acronym: FESSPRD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Michał Stasiowski, Principal Investigator, 2Department of Anaesthesiology and Intensive Therapy, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SilesianMUKOAiIT9
Record Dates: First submitted 2018-01-05; First posted 2018-01-31 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Endoscopic Sinus Surgery
Keywords: Pupillary Dilatation Reflex (PRD); Intraoperative Blood Loss (IBL); Boezaart Bleeding Scale (BBS); Spectral Entropy (SE); Adequacy of Anaesthesia (AoA); Total Intravenous Anaesthesia (TIVA); Sevoflurane; Desflurane
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SEVOFLURANE INHALATIONAL ANAESTHESIA (Experimental): concentration of sevoflurane in the exhalation gas will be maintained to ensure target SE between 40, remifentanyl solution will be administered intravenously at a rate 0,25 mcg/kg of body weight/minute, intraoperatively PRD measurement every 15 minutes; when PRD>5% infusion speed of remifentanyl will be increased by 50% every 5 minutes until PRD decreases below 5%
  Interventions: Drug: Remifentanil; Device: pupillary dilatation reflex
- DESFLURANE INHALATIONAL ANAESTHESIA (Experimental): concentration of desflurane in the exhalation gas will be maintained to ensure target SE 40, remifentanyl solution will be administered intravenously at a rate 0,25 mcg/kg of body weight/minute, intraoperatively PRD measurement every 15 minutes; when PRD>5% infusion speed of remifentanyl will be increased by 50% every 5 minutes until PRD decreases below 5%
  Interventions: Drug: Remifentanil; Device: pupillary dilatation reflex
- TIVA USING PROPOROL (Experimental): Infusion of propofol will be adjusted at target of SE 40,remifentanyl solution will be administered intravenously at a rate 0,25 mcg/kg of body weight/minute, intraoperatively PRD measurement every 15 minutes; when PRD>5% infusion speed of remifentanyl will be increased by 50% every 5 minutes until PRD decreases below 5%
  Interventions: Drug: Remifentanil; Device: pupillary dilatation reflex

INTERVENTIONS:
Drug: Remifentanil — a rate of infusion will be increased by 50% every 5 minutes until PRD decreases below 5%
  Other Names: Remifentanil infusion
Device: pupillary dilatation reflex — PRD value will me measured before the start of FESS after 5 minutes of remifentanyl infusion, when PRD sensitivity > 5% , infusion of remifentanyl will be increased by 50% until PRD sensitivity <5% and FESS will be started ; intraoperatively infusion of remifentanyl will be increased by 50% until PRD sensitivity <5%

SUMMARY:
The aim of this randomized trial is to assess the utility of Pupillary Dilatation Reflex (PRD) for monitoring pain perception intraoperatively and its influence on intraoperative blood loss, quality of surgical field using Boezaart Bleeding Scale (BBS) in patients undergoing functional sinus surgery (FESS) under total intravenous anaesthesia using propofol or volatile anaesthesia using sevoflurane or desflurane

DETAILED DESCRIPTION:
Intraoperative blood loss during FESS constitutes a major problem for a surgeon because it influences quality of surgical field. Each incident of haemorrhage makes the operator stop the procedure in order to bring back the optimal visualization of the intranasal anatomy. In the end it prolongs the time of procedure.

Currently, intraoperative blood loss is estimated based on Boezaart Bleeding Scale (BBS) (0 - no bleeding (cadaveric conditions), 1 - Slight bleeding, no suctioning required, 2 - Slight bleeding, occasional suctioning required, 3 - Slight bleeding, frequent suctioning required; bleeding threatens surgical field a few seconds after suction is removed, 4 - Moderate bleeding, frequent suctioning required, and bleeding threatens surgical field directly after suction is removed, 5 - Severe bleeding, constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely threatened and surgery usually not possible).

Recently, Pupillary Dilatation Reflex (PRD) was added as a surrogate variable showing the nociception-antinociception balance into above mentioned parameters constituting a novel approach in monitoring patients intraoperatively, known as adequacy of anaesthesia (AoA) or tailor-made anaesthesia. PRD value >5% reflects increased sensitivity to painful stimulus it constitutes the indication for administration of rescue analgesia intraoperatively.

This study aims at evaluating utility of PRD-directed analgesia using remifentanil on the intraoperative blood loss, haemodynamic stability and time duration of surgery in patients undergoing functional sinus surgery (FESS) under total intravenous anaesthesia using propofol or volatile anaesthesia using sevoflurane or desflurane Currently, FESS is most often performed using total intravenous anaesthesia (TIVA) which is by majority of anaesthesiologists believed to reduce the intraoperative blood loss compared to general anaesthesia using volatile anaesthetics, but current literature provides conflicting findings in this area if the sort of anaesthetic used influences quality of the surgical field.

ELIGIBILITY:
Inclusion Criteria:

* - written consent to participate in the study
* written consent to undergo functional endoscopic sinus surgery under general anaesthesia
* ASA (American Society of Anesthesiologists) I-III

Exclusion Criteria:

* age under 18 years old
* allergy to propofol
* pregnancy
* any anatomical malformation making PRD or SE measurement impossible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
blood loss postoperatively | end of operation,' assessment
  the investigators will measure the amount of blood loss in the suction bag in millilitres (ml) using a syringe after operation of FESS is completed

SECONDARY OUTCOMES:
heart rate stability intraoperatively | intraoperative assessment
  the investigators will measure heart rate during TIVAevery 5 minutes up to the end of the operation
PRD-guided pain perception intraoperatively | intraoperative assessment
  The investigators will measure PRD value and adjust infusion speed of remifentanyl, in the case of PRD value >5% the speed of remifentanyl infusion will accelerate by 50%, intraoperatively, every 15 minutes or at any change of BBS, up to the end of the operation
condition of surgical field | intraoperative assessment
  the surgeon will assess the quality of surgical field using BBS when the operation of FESS
total consumption of propofol | end of operation assessment
  The investigators will measure the consumption of propofol intraoperatively
total consumption of remifentanil | end of operation assessment
  The investigators will measure the consumption of remifentanyl intraoperatively
concentration of desflurane in end-expiratory gas | intraoperative assessment
  The investigators will measure theconcentration of desflurane in end-expiratory gas intraoperatively
concentration of sevoflurane in end-expiratory gas | intraoperative assessment
  The investigators will measure the concentration of sevoflurane in end-expiratory gas intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Przemysław Jałowiecki, Ph. Dr, Principal Investigator — Medical University of Silesia

IPD SHARING:
Plan to Share IPD: Yes
article in Laryngoscope in 2022, case reports
Supporting Information: ICF
Time Frame: starting 6 months after publication

REFERENCES:
- [Result] Cafiero T, Cavallo LM, Frangiosa A, Burrelli R, Gargiulo G, Cappabianca P, de Divitiis E. Clinical comparison of remifentanil-sevoflurane vs. remifentanil-propofol for endoscopic endonasal transphenoidal surgery. Eur J Anaesthesiol. 2007 May;24(5):441-6. doi: 10.1017/S0265021506002080. Epub 2007 Mar 12. PMID 17376252
- [Result] Sivaci R, Yilmaz MD, Balci C, Erincler T, Unlu H. Comparison of propofol and sevoflurane anesthesia by means of blood loss during endoscopic sinus surgery. Saudi Med J. 2004 Dec;25(12):1995-8. PMID 15711683
- [Result] Bhat Pai RV, Badiger S, Sachidananda R, Basappaji SM, Shanbhag R, Rao R. Comparison of surgical conditions following premedication with oral clonidine versus oral diazepam for endoscopic sinus surgery: A randomized, double-blinded study. J Anaesthesiol Clin Pharmacol. 2016 Apr-Jun;32(2):250-6. doi: 10.4103/0970-9185.182112. PMID 27275059
- [Result] Marzban S, Haddadi S, Mahmoudi Nia H, Heidarzadeh A, Nemati S, Naderi Nabi B. Comparison of surgical conditions during propofol or isoflurane anesthesia for endoscopic sinus surgery. Anesth Pain Med. 2013 Sep;3(2):234-8. doi: 10.5812/aapm.9891. Epub 2013 Sep 1. PMID 24282774
- [Result] Cardesin A, Pontes C, Rosell R, Escamilla Y, Marco J, Escobar MJ, Bernal-Sprekelsen M. Hypotensive anaesthesia and bleeding during endoscopic sinus surgery: an observational study. Eur Arch Otorhinolaryngol. 2014 Jun;271(6):1505-11. doi: 10.1007/s00405-013-2700-0. Epub 2013 Sep 20. PMID 24052249
- [Result] Cardesin A, Pontes C, Rosell R, Escamilla Y, Marco J, Escobar MJ, Bernal-Sprekelsen M. A randomised double blind clinical trial to compare surgical field bleeding during endoscopic sinus surgery with clonidine-based or remifentanil-based hypotensive anaesthesia. Rhinology. 2015 Jun;53(2):107-15. doi: 10.4193/Rhino14.185. PMID 26030032
- [Result] Drozdowski A, Sieskiewicz A, Siemiatkowski A. [Reduction of intraoperative bleeding during functional endoscopic sinus surgery]. Anestezjol Intens Ter. 2011 Jan-Mar;43(1):45-50. Polish. PMID 21786531
- [Result] Shen PH, Weitzel EK, Lai JT, Wormald PJ, Ho CS. Intravenous esmolol infusion improves surgical fields during sevoflurane-anesthetized endoscopic sinus surgery: a double-blind, randomized, placebo-controlled trial. Am J Rhinol Allergy. 2011 Nov-Dec;25(6):e208-11. doi: 10.2500/ajra.2011.25.3701. PMID 22185726
- [Result] Gomez-Rivera F, Cattano D, Ramaswamy U, Patel CB, Altamirano A, Man LX, Luong A, Chen Z, Citardi MJ, Fakhri S. Pilot study comparing total intravenous anesthesia to inhalational anesthesia in endoscopic sinus surgery: novel approach of blood flow quantification. Ann Otol Rhinol Laryngol. 2012 Nov;121(11):725-32. doi: 10.1177/000348941212101105. PMID 23193905
- [Result] Nekhendzy V, Lemmens HJ, Vaughan WC, Hepworth EJ, Chiu AG, Church CA, Brock-Utne JG. The effect of deliberate hypercapnia and hypocapnia on intraoperative blood loss and quality of surgical field during functional endoscopic sinus surgery. Anesth Analg. 2007 Nov;105(5):1404-9, table of contents. doi: 10.1213/01.ane.0000282781.56025.52. PMID 17959973